CLINICAL TRIAL: NCT02798536
Title: A Phase I Study of the Mesothelin-Targeted Immunotoxin LMB-100 With or Without Nab-Paclitaxel (Abraxane) in Patients With Malignant Mesothelioma
Brief Title: Mesothelin-Targeted Immunotoxin LMB-100 in People With Malignant Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160127; 16-C-0127
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Mesothelioma
Keywords: Immunotoxin; Mesothelin; Targeted Therapy
MeSH Terms: conditions — Mesothelioma | interventions — LMB-100; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A1/LMB-100 dose escalation (closed) (Experimental): De-escalating doses of LMB-100 in up to 18 subjects
  Interventions: Drug: LMB-100
- A2/LMB-100 dose expansion (closed) (Experimental): Fixed dose of LMB-100 as determined in Arm A1 in up to 16 subjects
  Interventions: Drug: LMB-100
- B1/LMB-100+ nab- paclitaxel dose escalation (Experimental): De-escalating doses of LMB-100 + fixed dose of nab-paclitaxel in up to 12 subjects
  Interventions: Drug: LMB-100; Drug: nab-paclitaxel
- B2/LMB-100+ nab- paclitaxel dose expansion (Experimental): Fixed dose of LMB-100 as determined in Arm B1 + fixed dose of nab-paclitaxel in up to 16 subjects
  Interventions: Drug: LMB-100; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: LMB-100 — Administered intravenous (IV) on days 1, 3 and 5 of a 21 day cycle for up to 4 cycles (Arms A1 and A2) or 2 cycles (Arms B1 and B2)
Drug: nab-paclitaxel — Arms B1 and B2 only. Administered intravenous (IV) on days 1 and 8 of each 21 day cycle for up to 6 cycles
  Arms: B1/LMB-100+ nab- paclitaxel dose escalation; B2/LMB-100+ nab- paclitaxel dose expansion

SUMMARY:
Background:

LMB-100 is a man-made protein. It is attracted to the mesothelin protein. This is found in many tumors, including mesothelioma. But it is found in only a very small number of normal tissues. After binding to mesothelin on tumors, LMB-100 attacks and kills cancer cells. Researchers want to test LMB-100 in people with advanced mesothelioma.

Objective:

To find a safe dose and anti-tumor activity of LMB-100 for people with advanced mesothelioma.

Eligibility:

Adults ages 18 and older with:

Advanced pleural or peritoneal mesothelioma that has not responded to platinum-based

therapy

Adequate organ function

Design:

Participants will be screened with:

Samples of tumor tissue or tumor fluid. These can be new or from a previous procedure.

Medical history

Physical exam

Blood, urine, and heart tests

Chest x-rays

Computed tomography (CT) or magnetic resonance imaging (MRI) scans

Fluorodeoxyglucose (FDG)-positron emission tomography (PET) scans

Participants will get LMB-100 on days 1, 3, and 5 of each 21-day cycle. It will be given through an intravenous (IV) catheter, a tube inserted in an arm vein. They will get standard medicines before each infusion to help prevent side effects. Each infusion lasts about 30 minutes. They will be monitored for up to 2 hours after.

During each cycle, participants will repeat the screening tests.

Participants will get the study drug for up to 4 cycles or until their disease worsens or they have intolerable side effects.

About 4-6 weeks after their last infusion, participants will have a follow-up visit. They will repeat the study tests.

Participants will have follow-up scans every 6 weeks until their disease gets worse.

Participants will be called about once a year to see how they are doing.

DETAILED DESCRIPTION:
Background:

* Although mesothelioma patients with a limited tumor burden may benefit from surgical resection, most patients have advanced disease at diagnosis and are not candidates for cytoreductive surgery.
* For mesothelioma patients who are not eligible for curative surgery, the median survival with supportive care alone is 6 months whereas with the current standard treatment, a combination of cisplatin and pemetrexed, the median survival is 12 months.
* Mesothelin, a tumor differentiation antigen, is expressed in over 95% of epitheloid mesothelioma. Mesothelin is a suitable candidate for targeted therapy due to its very limited expression in normal human tissue and its high expression in several tumors including mesothelioma.
* LMB-100 is a novel recombinant anti-mesothelin immunotoxin developed for the treatment of patients with solid tumors that express mesothelin. Mesothelin is targeted by linking a humanized fragment of the anti-mesothelin Fab to a de-immunized Pseudomonas exotoxin (PE).
* The clinical use of first generation immunotoxins such as SS1P was hampered mainly by their high immunogenicity. LMB-100 is a next generation PE-fusion protein that has been protein-engineered to maximally reduce its immunogenicity. LMB-100 has shown broad activity against different mesothelin expressing cancer cell lines and tumor xenograft models.

Objectives: Phase 1

To identify the recommended phase 2 dose (RP2D) of LMB-100 in patients with treatment refractory advanced epithelioid or biphasic mesothelioma and evaluate potential efficacy of the identified RP2D.

-Phase 2

To determine the efficacy of LMB-100 with respect to objective response rate in patients with treatment refractory advanced epithelioid or biphasic mesothelioma.

Eligibility:

* Age greater than or equal to 18 years
* Histologically confirmed advanced pleural or peritoneal mesothelioma
* Subjects must have had at least 1 prior chemotherapy regimen with last dose of previous therapy occurring at 3 weeks before the start of study treatment
* Adequate organ function
* Participants with central nervous system (CNS) metastases or prior pneumonectomy are excluded

Design:

* This is a Phase I, open-label study to evaluate the safety, pharmacokinetics, and activity of LMB-100 in patients with treatment refractory advanced epithelioid or biphasic mesothelioma.
* LMB-100 will be administered intravenously on days 1, 3 and 5 of each 21 day cycle for up to 4 cycles
* Tumor response will be assessed after every 2 cycles
* Optional tumor biopsies may be collected at baseline and after 2 cycles of therapy
* The accrual ceiling will be set at 30

ELIGIBILITY:
* INCLUSION CRITERIA (All Cohorts):
* Histologically confirmed epithelial or biphasic mesothelioma not amenable to potentially curative surgical resection. However, patients with biphasic tumors that have a more than or equal to 50% sarcomatoid component will be excluded. The diagnosis will be confirmed by the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI).
* Archival sample or fresh biopsy or tumor effusion must be available for confirmation of diagnosis.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to10 mm with spiral computed tomography (CT) scan.
* Patients must have had at least one prior chemotherapy regimen that includes pemetrexed and cisplatin or carboplatin. There is no limit to the number of prior chemotherapy regimens received.
* The last dose of previous therapy must have occurred at least 3 weeks prior to the start of study therapy. Palliative radiotherapy is allowed up to 2 weeks before the first LMB-100 infusion.
* Patients for whom no standard curable therapy exists
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of LMB-100 in patients <18 years of age, children are excluded from this study
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade less than or equal to 1, except alopecia (any grade) and Grade 2 peripheral neuropathy.
* Eastern Cooperative Oncology (ECOG) performance status (PS) 0 or1
* Adequate hematological function: neutrophil count of more than of equal to 1.5x10^9 cells/L, platelet count of greater than or equal to 100,000/microl, (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample) hemoglobin more than or equal to 9 g/dL
* Adequate Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 X upper limit of normal alkaline phosphate less than 2.5 X upper limit of normal unless bone metastasis is present (less than 5 X upper limit of normal) in the absence of liver metastasis.
* Bilirubin less than or equal to 1.5 mg/dL (excluding Gilbert's Syndrome, see below).
* Patients with Gilbert's syndrome will be eligible for the study. The diagnosis of Gilbert's syndrome is suspected in people who have persistent, slightly elevated levels of unconjugated bilirubin without any other apparent cause. A diagnosis of Gilbert's syndrome will be based on the exclusion of other diseases based on the following criteria:

  * Unconjugated hyperbilirubinemia noted on several occasions
  * No evidence of hemolysis (normal hemoglobin, reticulocyte count, and lactate dehydrogenase (LDH)
  * Normal liver function tests
  * Absence of other diseases associated with unconjugated hyperbilirubinemia
* Adequate renal function: creatinine less than 1.5 mg/dL OR creatinine clearance (by Cockcroft Gault formula) greater than or equal to 50 mL/min.
* Must have serum albumin > 2.5 mg/dL without intravenous supplementation
* Must have left ventricular ejection fraction > 50%
* Must have an ambulatory oxygen saturation of > 90% on room air
* Women of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or; (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

  * Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study therapy (including dose interruptions), while on study medication and for 3 months after the last dose of study therapy; and
  * Have a negative serum pregnancy test (<= -human chorionic gonadotropin (hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
* Men must agree to practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following discontinuation of study therapy, even if he has undergone a successful vasectomy.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA (All Cohorts):

-Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases. History or clinical evidence of CNS metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days.

Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant pulmonary disease other than primary cancer, uncontrolled diabetes mellitus, and/or significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina, or clinically significant pericardial effusion)

* Active or uncontrolled infections.
* Human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. HIV positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.
* Patients with prior pneumonectomy
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury greater than or equal to 28 days prior to the first LMB-100 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Dementia or altered mental status that would prohibit informed consent
* Live attenuated vaccinations 14 days prior to treatment
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100, breastfeeding should be discontinued if the mother is treated with LMB-100. These potential risks may also apply to other agents used in this study.
* Known hypersensitivity to any of the components of LMB-100
* High doses of systemic corticosteroids within 7 days prior to first dosing. High dose is considered as > 20 mg of dexamethasone a day (or equivalent) for > 7 consecutive days.

EXCLUSION CRITERIA (Cohort B only)

* Subjects must not have received paclitaxel nor nab-paclitaxel within 4 months prior to initiation of study therapy.
* Participants with contra-indication and/or history of sever hypersensitivity reactions to nab-paclitaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data in Biomedical Translational Research Information System (BTRIS) will be shared throughout the course of the study and indefinitely with the permission of the investigator.
Access Criteria: Clinical individual participant data (IPD) will be shared through the Biomedical Translational Research Information System (BTRIS) database for open ended analysis. All BTRIS subscribers, generally limited to the National Institutes of Health (NIH) Clinical Center, may request data.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0127.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 170mcg LMB-100: Dose Level 1: 170mcg LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 4 cycles.
- Dose Level -1: 140mcg LMB-100: Dose Level -1: 140mcg LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 4 cycles.
- Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel: Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel given intravenously. LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 2 cycles. Nab-Paclitaxel given intravenously on days 1 and 8 of each 21 day cycle for up to 6 cycles.
Period: Overall Study
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Started | 3 | 7 | 11
Completed | 3 | 7 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel | Total
Number analyzed (Participants) | 3 | 7 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 10 | 15
  >=65 years | 2 | 3 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.77 (19.07) | 57.09 (11.84) | 52.45 (16.46) | 54.9 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6 | 12
  Male | 2 | 2 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 7 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 6 | 8 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of LMB100 + Nab-paclitaxel
Description: Highest administered dose of LMB-100 + nab-paclitaxel at which no more than 1 of 6 participants experiences a dose limiting toxicity (DLT). A DLT is any of the following events attributed to LMB-100 and occurring within 21 days after the first dose of LMB-100 such as Grade 4 neutropenia, Grade 3 and 4 febrile neutropenia, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia associated with bleeding episodes. Grade ≥ 3 non-hematological toxicity with the exception of alopecia (any grade), Grade 3 nausea and vomiting without appropriate treatment, Grade 3 diarrhea lasting for ≤ 2 days with no fever or dehydration.
Time Frame: 3 weeks after initial dose
Population: Number of participants in the recommended Phase 2 (RP2D) of LMB-100 and the recommended Phase 2 Dose (RP2D) of LMB100 + Nab-paclitaxel are noted below.
Measure: Number; unit: mcg
Groups:
- All Participants: Dose Level 1: 170mcg LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 4 cycles.
  Dose Level -1: 140mcg LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 4 cycles.
  Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel given intravenously. LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 2 cycles. Nab-Paclitaxel given intravenously on days 1 and 8 of each 21 day cycle for up to 6 cycles.
Arm/Group | All Participants
Number analyzed (Participants) | 21
mcg
  Recommended Phase 2 (RP2D) of LMB-100: number analyzed (Participants) | 10
  Recommended Phase 2 (RP2D) of LMB-100 | 140
  Recommended Phase 2 Dose (RP2D) of LMB100 + Nab-paclitaxel: number analyzed (Participants) | 11
  Recommended Phase 2 Dose (RP2D) of LMB100 + Nab-paclitaxel | 100

2. Secondary Outcome: Number of Participants at Recommended Phase 2 Dose (RP2D) With Partial or Complete Response by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of participants at maximum tolerated dose (MTD) with partial or complete response measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: End of treatment, an average of 57.6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 7 | 11
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: At progression, up to 3.6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
months | 2.7 [2.7 to 3.0] | 2.7 [1.5 to 3.2] | 2.7 [1.3 to 3.6]

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS is defined as the duration of time from start of treatment to time of death.
Time Frame: At death, up to 60.8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
months | 33.5 [27.7 to 34.6] | 16.9 [6.8 to 60.8] | 10.1 [3.7 to 30.9]

5. Secondary Outcome: Number of Participants With LMB-100 Maximum Observed Serum Concentration (Cmax) of >100ng/mL
Description: Number of participants with LMB-100 Maximum observed serum concentration (Cmax) of >100ng/mL was measured by
Time Frame: Cycle 1 and Cycle 2 (each cycle is 21 days), approximately 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
Participants
  Cycle 1 | 3 | 7 | 10
  Cycle 2 | 2 | 4 | 3

6. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) Formation to LMB-100
Description: ADAs formation to LMB-100 were measured by the enzyme-linked immunosorbent assay (ELISA). The presence of ADAs (i.e., positive) may indicate the participant may have poor blood levels.
Time Frame: Cycle 1 and Cycle 2 (each cycle is 21 days), approximately 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 10
Participants
  Cycle 1 | 0 | 2 | 3
  Cycle 2 | 3 | 5 | 5
  No ADA formation | 0 | 0 | 2

7. Secondary Outcome: Number of Grade 3-5 Adverse Events Possibly, Probably, and/or Definitely Related to the LMB-100 +/- Nab-Paclitaxel
Description: Adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is serious, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 30 days after treatment
Measure: Number; unit: adverse events
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
adverse events
  Grade 3 hyponatremia possibly related | 0 | 0 | 1
  Grade 3 edema limbs possibly related | 0 | 0 | 1
  Grade 3 hypotension probably related | 0 | 0 | 1
  Grade 3 CPK increased probably related | 0 | 0 | 1
  Grade 3 atrial fibrillation probably related | 0 | 0 | 1
  Grade 3 hypoalbuminemia definitely related | 0 | 0 | 4
  Grade 3 hyponatremia definitely related | 0 | 2 | 0
  Grade 4 CPK increased probably related | 0 | 0 | 1

8. Secondary Outcome: Duration of Response (DOR)
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Progressive disease was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented by computed tomography (CT) scans performed every 6 weeks.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
months | NA [NA to NA] — Criteria not met for CR or PR so DOR not calculated, data is not available. | NA [NA to NA] — Criteria not met for CR or PR so DOR not calculated, data is not available. | NA [NA to NA] — Criteria not met for CR or PR so DOR not calculated, data is not available.

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 19 days for Dose Level 1, 52 months for Dose Level -1, and 42 months and 3 days for Dose Level -2.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
Participants | 3 | 7 | 11

10. Other Pre Specified Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: A DLT is any of the following events attributed to LMB-100 and occurring within 21 days after the first dose of LMB-100 such as Grade 4 neutropenia, Grade 3 and 4 febrile neutropenia, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia associated with bleeding episodes. Grade ≥ 3 non-hematological toxicity with the exception of alopecia (any grade), Grade 3 nausea and vomiting without appropriate treatment, Grade 3 diarrhea lasting for ≤ 2 days with no fever or dehydration.
Time Frame: First 21 days after first dose of LMB-100
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level -2: 100mcg LMB-100 +Nab Paclitaxel: Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel given intravenously. LMB-100 given intravenously on days 1, 3 and 5 of a 21 day cycle for up to 2 cycles. Nab-Paclitaxel given intravenously on days 1 and 8 of each 21 day cycle for up to 6 cycles.
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 +Nab Paclitaxel
Number analyzed (Participants) | 3 | 7 | 11
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 19 days for Dose Level 1, 52 months for Dose Level -1, and 42 months and 3 days for Dose Level -2.
Arm/Group | Dose Level 1: 170mcg LMB-100 | Dose Level -1: 140mcg LMB-100 | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/7 | 11/11
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/7 | 4/11
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 170mcg LMB-100 (N=3) | Dose Level -1: 140mcg LMB-100 (N=7) | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel (N=11)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Creatine phosphokinase (CPK) increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 170mcg LMB-100 (N=3) | Dose Level -1: 140mcg LMB-100 (N=7) | Dose Level -2: 100mcg LMB-100 + Nab-Paclitaxel (N=11)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (5) | 3 (8) | 4 (13)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (6) | 4 (10)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 3 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 2 (6) | 4 (22) | 9 (32)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 5 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 5 (9) | 6 (15)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 1 (1) | 1 (4)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (5) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (6)
Creatinine increased (Investigations) | 3 (18) | 3 (5) | 5 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) | 2 (3)
Ear and labyrinth disorders - Other, right ear clogging (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 3 (5) | 6 (9) | 9 (15)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Eye disorders - Other, Itching (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 5 (10) | 7 (9)
Fever (General disorders) | 1 (8) | 3 (19) | 3 (5)
Flushing (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, Peripheral intravenous(IV) infiltrated (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (8) | 4 (8) | 2 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, Blood lactate dehydrogenase increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (15) | 7 (18) | 5 (17)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 4 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (19) | 7 (35) | 10 (75)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (8)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 4 (10) | 9 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (11)
Hypotension (Vascular disorders) | 1 (1) | 4 (10) | 4 (6)
Infections and infestations - Other, Thrush (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Infusion related reaction (General disorders) | 0 (0) | 5 (8) | 2 (3)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Localized edema (General disorders) | 0 (0) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 3 (14) | 7 (34) | 11 (56)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (7) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (8) | 3 (7)
Pain (General disorders) | 1 (2) | 3 (6) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4)
Phlebitis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 1 (3) | 1 (2) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 3 (4) | 6 (16)
Skin and subcutaneous tissue disorders - Other, Decubitus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (7)
Weight gain (Investigations) | 2 (4) | 4 (5) | 6 (13)
Weight loss (Investigations) | 2 (4) | 0 (0) | 1 (4)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02798536/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT02798536/ICF_001.pdf